CLINICAL TRIAL: NCT00001062
Title: A Phase I Study of a Fixed-Schedule Regimen of Alternating Oral and Intravenous Ganciclovir for Treatment of Cytomegalovirus Retinitis
Brief Title: A Study of Ganciclovir in the Treatment of Cytomegalovirus of the Eyes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 278; 11254 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Infusions, Intravenous; Ganciclovir; Administration, Oral; Acquired Immunodeficiency Syndrome; Antiviral Agents; Cytomegalovirus Retinitis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To determine whether alternating oral ganciclovir with intravenous ( IV ) ganciclovir can prevent relapse of Cytomegalovirus ( CMV ) retinitis and improve quality of life in AIDS patients.

A systemic treatment strategy for CMV retinitis is needed that will be effective yet convenient to administer, without the need for a permanent indwelling IV catheter. Although oral ganciclovir has been used as maintenance following induction with IV ganciclovir, patients with reactivation of disease must be reinduced IV. A fixed-schedule regimen in which oral and IV ganciclovir are alternated may prevent reactivation and progression of disease, as opposed to the current therapeutic strategy in which changes in therapy are event-driven. Also, the duration of intermittent IV therapy required to control disease may be short enough to eliminate the need for an indwelling catheter.

DETAILED DESCRIPTION:
A systemic treatment strategy for CMV retinitis is needed that will be effective yet convenient to administer, without the need for a permanent indwelling IV catheter. Although oral ganciclovir has been used as maintenance following induction with IV ganciclovir, patients with reactivation of disease must be reinduced IV. A fixed-schedule regimen in which oral and IV ganciclovir are alternated may prevent reactivation and progression of disease, as opposed to the current therapeutic strategy in which changes in therapy are event-driven. Also, the duration of intermittent IV therapy required to control disease may be short enough to eliminate the need for an indwelling catheter.

Patients receive IV induction with ganciclovir for 2 weeks followed by an alternating course of 3 weeks of oral ganciclovir and 1 week of IV drug for four cycles (16 weeks). If CMV retinitis fails to arrest after initial induction, IV ganciclovir is administered for an additional 2 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Erythropoietin, G-CSF, or GM-CSF.
* Antiretrovirals.

Patients must have:

* HIV infection.
* Evaluable CMV retinitis with photographable lesions.
* Life expectancy of at least 6 months.
* No active AIDS-defining opportunistic infections or malignancies that require nephrotoxic or myelosuppressive therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Evidence of retinal vascular or related infectious disease or other retinal lesions that would interfere with the ability to detect responses to therapy or progression.
* Corneal, lens, or vitreous opacification precluding funduscopic exam.
* Clinically significant pulmonary or neurologic impairment other than seizure disorder or CNS mass lesion.
* Inability to obtain temporary IV access.
* Requirement for permanent catheters for IV ganciclovir administration.
* Uncontrolled diarrhea or nausea preventing ingestion of medicine.
* Known hypersensitivity to IV or oral ganciclovir.

Concurrent Medication:

Excluded:

* Immunomodulators.
* Biologic response modifiers.
* Interferon.
* Related investigational agents.
* CMV prophylaxis.
* Systemic acyclovir.
* Any nephrotoxic agent.
* Any concomitant therapy that would prohibit use of ganciclovir.

Prior Medication:

Excluded:

* Prior treatment for CMV retinitis.
* More than 4 months of prior ganciclovir or foscarnet, or within 4 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Study Completion 1998-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holland GN, Study Chair; Hardy WD, Study Chair
Locations (6):
- United States (6):
  - UCLA CARE Center CRS, Los Angeles, California
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Cornell University A2201, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Danner SA, Matheron S. Cytomegalovirus retinitis in AIDS patients: a comparative study of intravenous and oral ganciclovir as maintenance therapy. AIDS. 1996 Dec;10 Suppl 4:S7-11. PMID 9110064